CLINICAL TRIAL: NCT06238401
Title: An Open-label, Multi-center, Dose-escalation and Cohort Expansion Phase I/IIa Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile and Efficacy of ACR246 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Adcoris Biopharmacy Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACR246-101
Record Dates: First submitted 2024-01-17; First posted 2024-02-02 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACR246 for injection (Experimental): Administered by intravenous infusion on Day 1 every 3 weeks (Q3W).
  Interventions: Drug: ACR246 for injection

INTERVENTIONS:
Drug: ACR246 for injection — 80 mg/vial

SUMMARY:
The goal of the study is to evaluate the safety and tolerability of ACR246 in patients with advanced solid tumors, to determine the maximum tolerated dose (MTD) and Phase II recommended dose (RP2D) of ACR246.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be enrolled in this study:

1. Be willing to sign the ICF, be able to understand the study, and be willing to follow and be able to complete all the study procedures;
2. Male and female, aged 18 to 75 years (inclusive);
3. For phase I dose escalation study: Patients with histologically or cytologically confirmed recurrent or metastatic unresectable advanced solid tumors who experience disease progression after receiving systemic standard therapy, or have no standard therapy;
4. For phase IIa cohort escalation study: Patients with histologically or cytologically confirmed recurrent or metastatic unresectable advanced solid tumors who experience disease progression after receiving systemic standard therapy, or have no standard therapy, including the following malignant tumors:

   1. Esophageal cancer: Patients who experience disease progression after receiving prior ≥2 lines of chemotherapy;
   2. Colorectal cancer: Patients who experience disease progression after receiving prior ≥2 lines of chemotherapy;
   3. NSCLC: Patients with NSCLC meet the following conditions, and are unable to continue subsequent standard of care or have no standard of care available as judged by the investigator:

   i. Positive for driver genes (such as EGFR, ALK, ROS1, MET); disease progression after current standard targeted therapy; ii. Negative for driver genes (such as EGFR, ALK, ROS1, MET); disease progression after prior ≥1 line(s) of therapy, and use of platinum-based drugs in at least one regimen; d) Ovarian cancer: Patients who experience disease progression after receiving at least one prior line of chemotherapy; the patient must receive prior treatment with PARP inhibitors if harboring BRCA 1/2 mutations; e) Prostate cancer: Patients with metastatic castration-resistant prostate cancer who receive at least one prior systemic therapy; f) Other solid tumors: Patients who experience disease progression after receiving prior standard of care, have no standard of care available, or are currently unsuitable to receive standard of care.
5. Positive for 5T4 expression as detected by the central laboratory (phase IIa only);
6. Phase I: Presence of at least one evaluable lesion by imaging as per RECIST v1.1; phase IIa: Presence of at least one measurable lesion by imaging as per RECIST v1.1. Lesions that are previously treated with radiotherapy cannot be considered target lesions unless the lesions have unequivocal progression;
7. Toxicity from prior antitumor therapies returned to Grade ≤1 as defined by NCI-CTCAE v5.0, but with the exception for alopecia- or antitumor therapy-associated events that can be tolerated by patients as judged by the investigator;
8. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤1;
9. Adequate bone marrow, liver, kidney, and coagulation functions (refer to the upper limit of normal [ULN] of each clinical study site):

   Bone marrow (did not receive blood transfusion or use drugs that increase white blood cells and platelets, e.g., cytokines or erythropoietin, within 2 weeks prior to laboratory tests):

   Absolute neutrophil count (ANC) count ≥1.5×109/L; Platelet (PLT) ≥100×109/L; Haemoglobin (Hb) ≥90 g/L;

   Liver function:

   Total bilirubin (TBiL) ≤1.5 × ULN; ALT, AST ≤2.5 × ULN in patients without metastases to liver; ALT, AST ≤5 × ULN in patients with metastases to liver;

   Kidney function:

   Creatinine ≤1.5 × ULN or creatinine clearance (Ccr) ≥60 mL/min (according to the Cockcroft-Gault formula);

   Coagulation function:

   International normalized ratio (INR) ≤1.5 × ULN; Activated partial thromboplastin time (APTT) ≤1.5 × ULN;
10. Expected survival ≥3 months;
11. At rest, left ventricular ejection fraction (LVEF) ≥50%;
12. Eligible male patients of reproductive potential and female patients of childbearing potential, along with his/her partner, must agree to use medically acceptable contraceptive measures (e.g., hormonal contraception, barrier method, or abstinence, etc.) during the study and for at least 6 months after the last dose.

Exclusion Criteria:

Patients meeting any of the following criteria should be excluded from the study:

1. Comorbid with other primary malignant tumors, except for:

   1. Resolved non-invasive basal cell carcinoma or squamous cell carcinoma, and cervical carcinoma in situ;
   2. Or other malignant tumors with a more than 5-year disease free survival;
   3. Malignant tumors other than those with a more than 5-year disease free survival, but the patient may obtain benefits after enrollment as he/she has a stable condition assessed by the investigator (for phase I dose escalation study only);
2. Received any systemic antitumor therapies (including chemotherapy, radiotherapy, biological therapy, immunotherapy, etc.) within 4 weeks prior to the first dose of the investigational drug; Received small molecule targeted drugs, Chinese herbal medicines or Chinese patent medicines with antitumor indications or systemic immunomodulators (including but not limited to interferon, interleukin-2, and tumor necrosis factor) within 2 weeks prior to the first dose of the investigational drug;
3. Prior treatment with any 5T4-targeted drug therapy;
4. Presence of active brain metastases or spinal cord metastases, being ineligible for inclusion in the study as assessed by the investigator; however, patients who require no radiotherapy, surgery or treatment with corticosteroids to control the symptoms of metastases within 1 month prior to screening may be included in the study; patients with metastases to meninges will be excluded;
5. Known hypersensitivity to any of the active ingredients or excipients of ACR246, or documented history of allergy to protein drugs, experienced other serious allergic reactions, for which, the patient is not suitable to receive ACR246 as assessed by the investigator;
6. History of severe heart disease as assessed by the investigator, e.g., symptomatic cardiac failure congestive (CHF) [Class ≥2 as per New York Heart Association (NYHA) functional classification], and history of myocardial infarction or unstable angina pectoris within 6 months prior to screening;
7. Serious arrhythmia requiring medication, e.g., corrected QT interval (Frederica formula) >450 msec for male or >470 msec for female, complete left bundle branch block, third-degree atrioventricular block;
8. Uncontrolled hypertension after medication treatment (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg);
9. Dyspnoea at rest, severe primary pulmonary disorder currently requiring continuous oxygen therapy, history of interstitial lung disease and radiation pneumonitis, uncontrolled or potential risk of pulmonary fibrosis, or clinically active lung diseases as indicated by any proof;
10. Serious or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, heart, liver or kidney diseases), as assessed by the investigator;
11. Positive antibody tests for active hepatitis B (hepatitis B surface antigen positive and HBV DNA≥1×103 IU/mL), active hepatitis C (hepatitis C antibody positive and HCV RNA > lower limit of detection), active syphilis (treponema pallidum antibody positive and Rapid Plasma Reagin (RPR) titer positive), and human immunodeficiency virus (HIV) antibody positive, or any uncontrolled infections;
12. Had a major surgery or serious traumatic injuries (without complete recovery as assessed by the investigator) within 4 weeks prior to the first dose of the investigational drug, or plans to undergo a major surgery during the study;
13. Pregnant or lactating women;
14. Serious arterial/venous thrombosis (e.g., cerebrovascular accident [including transient ischaemic attack]), deep venous thrombosis, pulmonary embolism within 1 year prior to treatment with the investigational drug, or haemorrhagic diathesis within 30 days prior to enrollment, or existence of risks of massive gastrointestinal hemorrhage, as assessed by the investigator;
15. Use of strong cytochrome P450 3A enzymes (CYP450 3A) inhibitors or inducers could not be stopped during treatment with the investigational drug;
16. Active eye disorders, such as keratitis, corneal disorder or eye infection, requiring intervention (including surgery or drug therapy, etc.);
17. Other condition that in the opinion of the investigator is not suitable for the study, e.g., poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability: | 21days
  Incidence and characteristics of adverse events (AEs), serious adverse events (SAEs) and dose-limiting toxicities (DLTs).

SECONDARY OUTCOMES:
PK parameters of ACR246（Cmax） | 21days
  To assess the pharmacokinetic profile in patients with advanced solid tumors
PK parameters of ACR246（Tmax） | 21days
  To assess the pharmacokinetic profile in patients with advanced solid tumors
PK parameters of ACR246（t1/2） | 21days
  To assess the pharmacokinetic profile in patients with advanced solid tumors
PK parameters of ACR246（AUC0-t） | 21days
  To assess the pharmacokinetic profile in patients with advanced solid tumors
PK parameters of ACR246（AUC0-∞） | 21days
  To assess the pharmacokinetic profile in patients with advanced solid tumors
PK parameters of ACR246（CL） | 21days
  To assess the pharmacokinetic profile in patients with advanced solid tumors
PK parameters of ACR246（Vd） | 21days
  To assess the pharmacokinetic profile in patients with advanced solid tumors
PK parameters of ACR246（mean residence time (MRT)） | 21days
  To assess the pharmacokinetic profile in patients with advanced solid tumors

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Tumor Hospital, Beijing, Beijing Municipality
  - Zhejiang Cancer Hospital, Zhejiang, Hangzhou
  - Shandong First Medical University affiliated Cancer Hospital of Shandong, Shandong, Jinan
  - ShangHai Chest Hospital, Shanghai, Shanghai Municipality
  - ShangHai Sixth People's Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No